CLINICAL TRIAL: NCT04228939
Title: Therapist-guided Smartphone-based Aftercare for Inpatients With Severe Anorexia Nervosa (SMART-AN): a Randomized Controlled Trial
Brief Title: Smartphone-based Aftercare for Inpatients With Anorexia Nervosa
Acronym: SMART-AN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Schoen Clinic Roseneck (Unknown); Swiss Anorexia Nervosa Foundation (Unknown)
Responsible Party: Principal Investigator, Schlegl Sandra, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 78-17
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental)
  Interventions: Behavioral: Recovery Record aftercare
- Control group (CG) (Active Comparator)
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Recovery Record aftercare — Patients randomized to IG receive a therapist-guided smartphone-based aftercare intervention for a period of 16 weeks. The patients are invited to download for free the German version of "Recovery Record" at the App Store (iPhone) or the Google Play Store (android) to their smartphone and to link with the aftercare therapist. After discharge, patients are asked to monitor their meals at least three times per day (breakfast, lunch, and dinner), that is, to produce a minimum of three logs per day over the subsequent 16 weeks. Furthermore, patients are instructed to monitor their thoughts and feelings as well as their (disordered) behaviors. The aftercare therapist also sets the patients clinical post-discharge goals and makes coping skill suggestions. Individual therapist feedback is provided in-app twice per week during the first four weeks, once per week in weeks 4-8, every other week in weeks 8-12 and once in week 16.
  Arms: Intervention group (IG)
Behavioral: Treatment as usual (TAU) — Patients randomized to CG receive TAU i.e. patients and their physicians or therapists decide on post-discharge treatment which is documented at T1 and T2.
  Arms: Control group (CG)

SUMMARY:
Inpatient treatment for patients with anorexia nervosa (AN) is recommended in extreme or severe cases after failure of outpatient treatment and is highly effective. However, a number of patients show symptom increase and relapse after discharge. The aim of this study is to evaluate the efficacy of a guided smartphone-based aftercare intervention following inpatient treatment of patients with AN to support symptom stabilization or continued improvement.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a severe, often chronic and life-threatening disorder. Relapse after treatment is common with relapse rates ranging between 9 and 52% and being highest within the first year following treatment particularly as early as 3 months posttreatment. Even if weight restoration is achieved, it is quite difficult for patients to sustain improvements after treatment, so aftercare and relapse prevention are essential research topics. There is a recent review on internet- and mobile-based aftercare and relapse prevention in mental disorders that concludes that there is some evidence that such interventions are feasible instruments for maintaining treatment gains for some mental disorders, including eating disorders (EDs). However, the authors claim for further high quality, large-scale trials that are needed to expand research fields. So, the aim of this study is to prove the efficacy of a guided smartphone-based aftercare intervention for inpatients with AN. Our primary hypothesis is that at the end of aftercare intervention (T1), the intervention group shows a significantly lower eating disorder symptomatology than the control group.

Eligible patients with AN who are discharged from inpatient treatment are randomized either to receive a 4-month smartphone-based aftercare intervention with therapist feedback as an add-on element to treatment as usual (TAU) or TAU alone. Assessments include structured interviews as well as online questionnaires and are taken at baseline (discharge, T0), end of the aftercare intervention (T1) as well as 6-month follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of AN (DSM-5: 307.1),
* sex: female,
* age: from 12 years onwards to 60 years,
* regular completion of inpatient treatment,
* at least a length of inpatient stay of 6 weeks,
* BMI at discharge at least 15, at least a 1-point BMI increase during inpatient treatment,
* owner of a smartphone,
* informed consent of the patient and, in case of minors, also of the parents.

Exclusion Criteria:

* major depression (BDI-II > 29 at discharge),
* suicidal tendency (item 9 of BDI-II > 1 at discharge),
* very high level of care after inpatient treatment (e.g. therapeutic living community, day clinic),
* pregnancy.

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Eating Disorder Severity (assessor-based) | Measured at baseline (discharge), at week 16 (end of treatment) and 6 month follow-up
  The Eating Disorder Examination (EDE) will be used to measure asessor-based eating disorder symptom severity over time.

SECONDARY OUTCOMES:
Changes in Body-Mass-Index (BMI) | Measured at baseline, week 16 and 6 month follow-up
  Weight and height will be used to measure BMI over time.
Changes in Eating Disorder Severity (self-report) | Measured at baseline, week 16 and 6 month follow-up
  The Eating Disorder Examination Questionnaire (EDE-Q) will be used to measure self-reported eating disorder symptom severity over time.
Changes in depressive symptoms | Measured at baseline, week 16 and 6 month follow-up
  The Beck Depression Inventory-II (BDI-II) will be used to measure depressive symptoms over time.
Changes in stages of change regarding specific eating disorder behaviors | Measured at baseline, week 16 and 6 month follow-up
  The Stages of Change Questionnaire for Eating Disorders (SOCQ-ED) will be used to measure changes in stages of change regarding specific eating disorder behaviors over time.
Changes in self-efficay | Measured at baseline, week 16 and 6 month follow-up
  The General Self-Efficacy Scale (GSE) will be used to measure self-efficacy over time.
Participant satisfaction with the app and the aftercare intervention | Measured at week 16
  A self-developed questionnaire will be used to assess self-reported satisfaction with the app and the aftercare intervention.
Additional outpatient and inpatient treatment after discharge | Measured at week 16 and 6 month follow-up
  Number and length of outpatient or inpatient treatment (rehospitalization) since discharge will be assessed.
Adherence to the smartphone-based aftercare intervention | Measured from baseline to week 16
  Adherence will be measured via dichotomous outcome of drop-out (individuals will be considered as drop-out if they fail to login to the app at all for a period of 14 consecutive days. Adherence will be assessed through application usage data.
Adherence to self-monitoring tasks | Measured from baseline to week 16
  Frequency of self-monitoring entries will be tracked automatically through the program server

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Schlegl, PhD, Principal Investigator — Ludwig Maximilian University Munich
Locations (1):
- Schoen Clinic Roseneck, Prien am Chiemsee, Germany

IPD SHARING:
Plan to Share IPD: No